CLINICAL TRIAL: NCT00814346
Title: Effect of Oral EGb761® on Brain Glucose Metabolism in Three Groups of Elderly With Memory Complaint, Mild Alzheimer's Disease, and Cognitively Normal Elderly. Phase II, Randomised, Double-blind, Parallel Groups, Placebo-controlled Study
Brief Title: Effect of EGb761® on Brain Glucose Metabolism in Three Groups of Elderly Defined by Cognitive Functions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2-39-00240-134; 2007-005377-63 (EudraCT Number)
Record Dates: First submitted 2008-12-23; First posted 2008-12-24 (Estimated); Results first posted 2016-03-28 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-01

CONDITIONS: Alzheimer's Disease; Cognitive Impairment
Keywords: Mild Alzheimer's disease (AD) patients; Memory complaint patients with cognitive impairment (MC); Memory complaint patients cognitively normal (CNE)
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Ginkgo biloba extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- EGb 120 mg (Active Comparator)
  Interventions: Drug: EGb761®
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EGb761® — Four weeks for AD patients, 18 months for MC and CNE patients
  Arms: EGb 120 mg
Drug: Placebo — Placebo 1 tablet BID
  Arms: Placebo

SUMMARY:
The aim of the study is to evaluate the effect of EGb761®, in comparison to placebo, on cerebral glucose metabolism, in three groups of elderly patients: newly diagnosed mild Alzheimer's disease (AD), memory complaint patients with cognitive impairment (MC) and memory complaint patients cognitively normal (CNE). The first phase includes four weeks treatment with EGb761® for all groups, with change in brain glucose metabolism at month 1 using 18 FDG-PET, as primary endpoint which will be followed by an open 17 months follow-up (FU) period with EGb761® treatment in MC and CNE patients.

ELIGIBILITY:
Inclusion Criteria:

* Group Specific Inclusion Criteria:

Cognitively normal elderly (CNE)

* Spontaneous memory complaint by patient,
* Mini-Mental State Exam score ≥ 28.
* Clinical Dementia Rating = 0.
* No Diagnostic And Statistical Manual Of Mental Disorders, Fourth Edition (DSMIV) criteria for Dementia.

Memory complaints (MC) :

* Spontaneous memory complaint by patient
* Mini-Mental State Exam score ≥ 25
* Clinical Dementia Rating 0.5.
* No DSMIV criteria for Dementia.

Mild Alzheimer's Disease (AD):

* Mini Mental Status Examination (MMSE) between 20 and 28 (inclusive).
* Clinical Dementia Rating ≥ 1.0
* DSMIV criteria for Dementia.
* National Institute of Neurological and Communicative Diseases and Stroke / Alzheimer's Disease and Related Disorders Association(NINCDS/ADRDA) criteria for probable AD.
* Newly diagnosed patients without treatment by Cholinesterase Inhibitors or Memantine.
* ≥ 65 years of age, both sex
* Geriatric Depression Scale (GDS) < 15
* Informed consent signed by the patient or, if necessary by legal representative

Exclusion Criteria:

* Contraindication to Magnetic Resonance Imaging (MRI) and/or Positron-Emission Tomography (PET) scan
* Forbidden Concomitant medications (Cholinesterase inhibitors and memantine, Specific psychoactive medications,e.g., neuroleptics, chronic anxiolytics including meprobamate, or sedative hypnotics other than benzodiazepines, Monoamine oxidase inhibitors (MAOIs) including selective MAOIs. Drugs acting on cerebral nervous system, Antidiabetes medications , Antioxidants medications, Medications known to interfere with cognitive evaluations
* Significant neurological disease and psychiatric disorders/psychotic feature
* Significant medical illness

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 49 (Actual)
Dates: Start 2008-10; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (8):
- France (8):
  - Hôpital Corentin Celton 4 parvis Corentin Celton, Issy-les-Moulineaux
  - Hôpital de Juvisy, Juvisy-sur-Orge
  - CMPI "Les Rives de Seine", Le Vésinet
  - Centre Hospitalier d'Orsay 4 place du Général Leclerc, Orsay
  - Private practice, Paris
  - Hôpital Broca 54-56 rue Pascal, Paris
  - Observatoire de l'âge, Paris
  - Hôpital Paul Brousse 12 av Paul-Vaillant-Couturier, Villejuif

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 63 participants were screened of which 49 subjects were randomised to either EGb761 and Placebo treatment groups (double-blind period).
  The 49 randomised subjects consisted of three groups of elderly subjects: Cognitively normal elderly (CNE), Memory Complaint (MC) and Alzheimer's Disease (AD).
Groups:
- EGb761 120 mg: EGb761 120 mg tablet twice a day for 4 weeks (Double-blind phase) for CNE, MC, and AD patients and 17 months (Open phase) for CNE and MC patients
- Placebo: Placebo 1 tablet twice a day for 4 weeks CNE, MC, and AD patients
Period: Double-blind Phase (4 Weeks)
Arm/Group | EGb761 120 mg | Placebo
Started | 23 | 26
CNE | 10 | 13
MC | 10 | 11
AD | 3 | 2
Completed | 23 | 23
Not Completed | 0 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Not otherwise specified | 0 | 2
Period: Open Phase (17 Months)
Arm/Group | EGb761 120 mg | Placebo
Started | 41 (Open period was treated with EGB761®. 41 subjects accepted follow-up open period(21 in CNE,20 in MC)) | 0 (This was an open period, without placebo arm, the number of subject on placebo is 0.)
CNE | 21 | 0
MC | 20 | 0
AD | 0 (Open period was not proposed to AD subjects.) | 0
Completed | 31 | 0
Not Completed | 10 | 0
Not completed — Adverse Event | 5 | 0
Not completed — Consent | 2 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Not otherwise specified | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EGb761 120 mg | Placebo | Total
Number analyzed (Participants) | 23 | 26 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.1 (6.2) | 76.6 (5.3) | 75.85 (5.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 32
  Male | 8 | 9 | 17
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.49 (4.46) | 25.03 (4.40) | 24.76 (4.43)
Educational Level [Number; unit: participants]
  Level 1: Primary only | 1 | 0 | 1
  Level 2: School certificate | 2 | 5 | 7
  Level 3: Completed secondary | 3 | 6 | 9
  Level 4: University | 17 | 15 | 32

OUTCOME MEASURES:

1. Secondary Outcome: Change in Brain Glucose Metabolism in the MC and CNE Groups
Description: Brain glucose metabolism measured by 18FDG PET
  SUVBSA2 = [Brain radioactivity (Bq/cc)] / [Injected dose (MBq)/BSA2] x [Blood glucose (g/l)]
  BSA2(m^2) = 0.007184 x Height (cm)^0.35 x weight (kg)^0.80
Time Frame: From Baseline (Month 0) to Month 18
Population: ITT population. N=Number of subjects with assessment.
Measure: Median (Full Range); unit: SUVBSA2
Groups:
- EGb 120 mg (Open Phase - CNE): EGb761 120 mg tablet twice a day for 17 months (open phase) for CNE patients
- EGb 120 mg (Open Phase - MC): EGb761 120 mg 17 months (open phase) for MC patients
Arm/Group | EGb 120 mg (Open Phase - CNE) | EGb 120 mg (Open Phase - MC)
Number analyzed (Participants) | 18 | 14
SUVBSA2
  Cerebellum | -0.07 [-0.3 to 0.1] | 0 [-0.5 to 0.2]
  Left cerebral cortex | -0.06 [-0.3 to 0.1] | -0.08 [-0.5 to 0.1]
  Left thalamus | -0.03 [-0.2 to 0.1] | -0.02 [-0.8 to 0.1]
  Left caudate nucleus | -0.11 [-0.8 to 0.2] | -0.01 [-0.6 to 0.2]
  Left putamen nucleus | 0.07 [-0.3 to 0.2] | 0.00 [-0.5 to 0.3]
  Left ventral striatum | -0.05 [-0.5 to 0.3] | -0.09 [-0.5 to 0.1]
  Left globus pallidus | 0.00 [-0.3 to 0.2] | -0.01 [-0.2 to 0.1]
  Right cerebral cortex | -0.07 [-0.3 to 0.1] | -0.06 [-0.3 to 0.1]
  Right thalamus | 0.04 [-0.3 to 0.2] | -0.00 [-0.9 to 0.2]
  Right caudate nucleus | 0.03 [-0.6 to 0.2] | -0.02 [-0.6 to 0.3]
  Right putamen nucleus | 0.04 [-0.5 to 0.2] | 0.02 [-0.3 to 0.3]
  Right ventral striatum | 0.01 [-0.4 to 0.3] | -0.05 [-0.6 to 0.4]
  Right globus pallidus | 0.06 [-0.3 to 0.4] | 0.06 [-0.2 to 0.6]

2. Secondary Outcome: Change in Cognitive Tests-Clinical Dementia Rating (CDR) Score in MC and CNE Groups
Description: CDR is a structured interview to collect information regarding subject's memory in a standard way from both the patient and the helper. Scores are calculated using below scale; q CDR=No dementia (score: 0), q CDR=Very mild dementia (score: 0.5), q CDR=Mild dementia (score: 1), q CDR=Moderate dementia (score: 2) and q CDR=Severe dementia (score: 3).
Time Frame: From Baseline (Month 0) to Month 9
Population: ITT population. N=Number of subjects with assessment.
Measure: Median (Full Range); unit: CDR overall score
Groups:
- EGb 120 mg (Open Phase - MC): EGb761 120 mg tablet twice a day for 17 months (open phase) for MC patient
Arm/Group | EGb 120 mg (Open Phase - CNE) | EGb 120 mg (Open Phase - MC)
Number analyzed (Participants) | 20 | 18
CDR overall score | 0.00 [0.0 to 0.5] | 0.00 [-0.5 to 0.5]

3. Secondary Outcome: Change in Cognitive Tests-Geriatric Depression Scale (GDS) Score in MC and CNE Groups
Description: The Geriatric Depression Scale is a self-administered depression scale, which was developed as a basic screening measure for depression in older adults. By "yes" or "no" answers, scores permit to classify patients into groups of "severely depressed" (score of 21 to 30), "moderately depressed" (score of 11 to 20) and "normal" (score of 0 to10). It takes10 to 15 minutes to administer.
Time Frame: From Baseline (Month 0) to Month 9
Population: ITT population. N=Number of subjects with assessment.
Measure: Median (Full Range); unit: GDS Score
Groups:
- EGb 120 mg (Open Phase - MC): EGb761 120 mg tablet twice a day for 17 months (open phase) for MC patients
Arm/Group | EGb 120 mg (Open Phase - CNE) | EGb 120 mg (Open Phase - MC)
Number analyzed (Participants) | 19 | 17
GDS Score | -2.00 [-6.0 to 8.0] | 0.00 [-5.0 to 9.0]

4. Secondary Outcome: Change in Cognitive Tests-Verbal Fluency in MC and CNE Groups
Description: Subjects completed a verbal fluency test. Higher scores represent higher levels of verbal fluency. Minimum score=0 and Maximum score= N/A.
  Letter fluency: this task consists of enouncing as many words as possible that begin with a given letter of the alphabet. Participants are not allowed to use proper names.
  Categorical fluency: in this task participants are asked to list as many words as possible that belong to a given semantic category (e.g. animals, fruits, towns) Each condition foresees 60 sec of word generation time. The score corresponds to the number of words correctly given. The verbal fluency task measures semantic storage and executive retrieval functions.
Time Frame: From Baseline (Month 0) to Month 9
Population: ITT population. N=Number of subjects with assessment.
Measure: Median (Full Range); unit: Number of good answers
Arm/Group | EGb 120 mg (Open Phase - CNE) | EGb 120 mg (Open Phase - MC)
Number analyzed (Participants) | 18 | 18
Number of good answers
  Categorical verbal fluency | -1.50 [-14.0 to 11.0] | -2.00 [-16.0 to 6.0]
  Lexical verbal fluency | -1.00 [-14.0 to 10.0] | 2.00 [-18.0 to 22.0]

5. Primary Outcome: Change in Brain Glucose Metabolism Measured Using 18-Fluorodeoxyglucose Positron Emission Tomography (18FDG-PET)
Description: Following statistical parametric mapping (SPM) analyses were performed by the Commissariat à l'Energie Atomique (CEA):
  * The comparison between treatment groups separately for each group of elderly subjects (CNE and MC groups only)
  * The comparison between the two groups of elderly subjects (CNE and MC groups only) by treatment group
  FDG PET demonstrates reductions in the cerebral glucose metabolism that may occur a few years before the overt clinical manifestation of disease.
  SUVBSA2 = [Brain radioactivity (Bq/cc)] / [Injected dose (MBq)/BSA2] x [Blood glucose (g/l)]
  BSA2(m^2) = 0.007184 x Height (cm)^0.35 x weight (kg)^0.80
  Standardized Uptake Value (SUV) Body Surface Area (BSA)
Time Frame: From Baseline (Month 0) to Week 4 (Month 1) - Double blind phase
Population: Intention to treat (ITT) population: All treated CNE and MC patients
Measure: Median (Full Range); unit: SUVBSA2
Groups:
- EGb761 120 mg (CNE); EGb761 120 mg (MC): EGb761 120 mg tablet twice a day for 4 weeks (Double-blind phase) for CNE, MC, and AD patients
- Placebo (CNE); Placebo (MC): Placebo 1 tablet twice a day for 4 weeks for CNE, MC and AD patients
Arm/Group | EGb761 120 mg (CNE) | Placebo (CNE) | EGb761 120 mg (MC) | Placebo (MC)
Number analyzed (Participants) | 10 | 11 | 10 | 10
SUVBSA2
  Cerebellum | -3.40 [-16.4 to 18.7] | -1.07 [-22.8 to 33.5] | -7.58 [-29.7 to 26.4] | -3.09 [-16.4 to 22.4]
  Left cerebral cortex | -8.56 [-14.0 to 22.0] | 2.25 [-28.9 to 35.9] | 0.44 [-36.3 to 35.8] | -0.32 [-33.9 to 30.7]
  Left thalamus | -8.46 [-23.3 to 25.1] | -0.06 [-39.6 to 37.4] | -2.09 [-35.2 to 30.1] | -6.19 [-38.9 to 31.2]
  Left caudate nucleus | -0.68 [-28.0 to 29.1] | 4.60 [-23.8 to 49.6] | 2.16 [-35.8 to 53.4] | 3.27 [-51.4 to 25.3]
  Left putamen nucleus | -1.91 [-23.7 to 26.3] | -0.19 [-23.5 to 55.8] | 2.15 [-46.0 to 46.2] | -6.20 [-49.1 to 39.8]
  Left ventral striatum | 1.49 [-53.5 to 19.7] | -7.29 [-30.4 to 67.5] | 2.37 [-22.3 to 24.4] | -4.62 [-53.8 to 33.8]
  Left globus pallidus | -4.33 [-26.3 to 19.4] | -1.26 [-9.4 to 39.2] | -7.75 [-28.5 to 14.0] | -8.72 [-24.7 to 26.3]
  Right cerebral cortex | -7.49 [-25.3 to 21.4] | 0.19 [-29.4 to 38.2] | -7.11 [-32.5 to 35.5] | -6.59 [-36.1 to 31.3]
  Right thalamus | -7.40 [-27.3 to 28.7] | -2.05 [-46.6 to 41.5] | -3.87 [-29.9 to 28.1] | -7.72 [-43.4 to 31.1]
  Right caudate nucleus | -1.59 [-36.2 to 29.1] | -0.66 [-23.7 to 46.0] | -9.21 [-34.2 to 40.9] | -6.45 [-41.3 to 16.7]
  Right putamen nucleus | -6.31 [-42.9 to 30.8] | -2.73 [-39.1 to 52.8] | -8.84 [-41.7 to 41.8] | -5.36 [-50.4 to 25.5]
  Right ventral striatum | -7.08 [-23.8 to 32.8] | -0.76 [-43.7 to 41.5] | -8.21 [-27.6 to 65.5] | -0.59 [-51.4 to 27.2]
  Right globus pallidus | -2.04 [-21.1 to 17.3] | -1.72 [-22.1 to 40.4] | -5.99 [-23.0 to 33.7] | -1.24 [-35.0 to 17.2]

6. Secondary Outcome: Change in Cognitive Tests-Mini Mental Status Examination (MMSE) Score in MC and CNE Groups
Description: MMSE is a brief screening instrument used to assess cognitive function in elderly participants. It assesses orientation, memory, attention, ability to name objects, follow verbal and written commands, write a sentence, and copy figures. Total score ranges from 0 to 30, with a lower score indicating greater disease severity.
Time Frame: From Baseline (Month 0) to Month 9
Population: ITT population. N=Number of subjects with assessment.
Measure: Median (Full Range); unit: MMSE Score
Arm/Group | EGb 120 mg (Open Phase - CNE) | EGb 120 mg (Open Phase - MC)
Number analyzed (Participants) | 19 | 18
MMSE Score | 0.00 [-2.0 to 1.0] | 0.00 [-6.0 to 4.0]

7. Secondary Outcome: Change in Cognitive Tests-Clock Drawing Test Score in MC and CNE Groups
Description: Clock drawing test is a visuo-constructive task, where subjects are asked to draw the face of a clock in a pre-drawn circle and then to draw in the arms to denote 16:45 (a quarter to five). The drawing can then be evaluated by a quantitative scoring method, which is based on the degree of completion of the drawing. The scoring system ranges from 0 to 6 with higher scores reflecting a greater number of errors and more impairment.
Time Frame: From Baseline (Month 0) to Month 9
Population: ITT population. N=Number of subjects with assessment.
Measure: Median (Full Range); unit: Clock drawing test score
Arm/Group | EGb 120 mg (Open Phase - CNE) | EGb 120 mg (Open Phase - MC)
Number analyzed (Participants) | 18 | 18
Clock drawing test score | 0.00 [-3.0 to 2.0] | 0.00 [-5.0 to 3.0]

8. Secondary Outcome: Change in Cognitive Tests-Cube Drawing Test Score in MC and CNE Groups
Description: Cube drawing: Subjects are asked to draw a cube by heart. In case of failure, a model of a cube is given to the subjects to copy.
  The score system ranges from 0 (worse score) to 6 (best score). Score calculation is following: 1 point by face with 4 sides, 2 points for each face where each angle should be respected.
Time Frame: From Baseline (Month 0) to Month 9
Population: ITT population. N=Number of subjects with assessment.
Measure: Median (Full Range); unit: Cube drawing test score
Arm/Group | EGb 120 mg (Open Phase - CNE) | EGb 120 mg (Open Phase - MC)
Number analyzed (Participants) | 18 | 18
Cube drawing test score | 0.00 [-2.0 to 1.0] | 0.00 [-4.0 to 5.0]

9. Secondary Outcome: Change in Cognitive Tests in MC and CNE Groups - Total Immediate Recall and Delayed Recall Scores of the Free and Cued Selective Reminding Test (FCSRT)
Description: Free and Cued Selective Reminding Test (FCSRT) Assessment of verbal episodic memory. By this test performances in free recalls, cued recalls and in a recognition task can be analysed, because the process of encoding is controlled.
  Subjects are asked to remember a list of 16 words. Three tasks of free and cued recalls, as well as one recognition task and one delayed recall give the scores.
  Total recall is obtained by the addition of cued recalls to free recalls. Maximum score is 48 for immediate: 16 words X 3 corresponding to immediate free recall + immediate cued recall + immediate recognition test.
  Maximum score is 64 (better score) when delayed recall : 16 words X 4 . The minimum score is 0 (worse).
Time Frame: From Baseline (Month 0) to Month 9
Population: ITT population. N=Number of subjects with assessment.
Measure: Median (Full Range); unit: Recall score
Arm/Group | EGb 120 mg (Open Phase - CNE) | EGb 120 mg (Open Phase - MC)
Number analyzed (Participants) | 18 | 18
Recall score
  Total Immediate Recall Score | 1.00 [-1.0 to 10.0] | 0.00 [-10.0 to 11.0]
  Total Delayed Recall Score | 0.00 [-4.0 to 6.0] | 0.00 [-4.0 to 5.0]

10. Secondary Outcome: Change in Cognitive Tests-Age-Adjusted Logical Memory (MEM III) in MC and CNE Groups
Description: Subjects are asked to memorize two short stories, one consisting of 24, the other one of 26 information units. After the stories have been read aloud by the investigator, subjects are asked to enounce all items of information they can remember (free recall). Correctly reported items are added for each story. This test applies analytical capacities, as well as auditive and verbal synthesis, working memory and episodic memory.
  Score range from 0(worst) to 75 (better).
Time Frame: From Baseline (Month 0) to Month 9
Population: ITT population. N=Number of subjects with assessment.
Measure: Median (Full Range); unit: Age adjusted score
Arm/Group | EGb 120 mg (Open Phase - CNE) | EGb 120 mg (Open Phase - MC)
Number analyzed (Participants) | 18 | 17
Age adjusted score | 1.00 [-5.0 to 6.0] | -1.00 [-4.0 to 7.0]

11. Secondary Outcome: Change in Cognitive Tests-Age-Adjusted Wechsler Adult Intelligence Scale (WAIS) in MC and CNE Groups
Description: Wechsler Adult Intelligence Scale (WAIS) In this test subjects are asked to say how two seemingly dissimilar items might in fact be similar (14 item couples). This test involves especially abstract thinking and concept capacities.
  Cognitive Tests-Age-Adjusted Wechsler Adult Intelligence Scale (WAIS): 19 tests on similarities. The items 1 to 5 are graded from 1 (good) to 0 (bad), and the items 6 to 19 are graded from 2 (good) to 0 (bad). Item 6 and 7 can be repeated. At the end, the worst total score is 0, the best total score is 33.
Time Frame: From Baseline (Month 0) to Month 9
Population: ITT population. N=Number of subjects with assessment.
Measure: Median (Full Range); unit: Age adjusted score
Arm/Group | EGb 120 mg (Open Phase - CNE) | EGb 120 mg (Open Phase - MC)
Number analyzed (Participants) | 17 | 18
Age adjusted score | 1.00 [-3.0 to 5.0] | 1.00 [-3.0 to 5.0]

12. Secondary Outcome: Change in Cognitive Tests-Time to Perform Trail Making Test (TMT) in MC and CNE Groups
Description: TMT is a neuropsychological test of visual attention and task switching. The task requires a subject to 'connect-the-dots' of 25 consecutive numbers (1,2,3,etc.) on a sheet of paper or computer screen. The goal of the subject is to finish the test as quickly as possible and the time taken to complete the test is used as the primary performance metric (in seconds). The maximum time allowed is 300 seconds. A negative change score indicates improvement.
  First, in the TMT A, the subject has to connect numbers increasingly as fast as possible.
  The TMT B requires the subject to connect and letters in an alternating pattern (1-A-2-B-3-C, etc.) in as little time as possible.
Time Frame: From Baseline (Month 0) to Month 9
Population: ITT population. N=Number of subjects with assessment.
Measure: Median (Full Range); unit: Seconds
Arm/Group | EGb 120 mg (Open Phase - CNE) | EGb 120 mg (Open Phase - MC)
Number analyzed (Participants) | 21 | 20
Seconds
  Task A (N=17,18) | 2.00 [-43.0 to 41.0] | 2.50 [-18.0 to 31.0]
  Task B (N=17,16) | 0.00 [-200.0 to 56.0] | -5.50 [-57.0 to 113.0]

13. Secondary Outcome: Number of Subjects Conversion to Alzheimer's Dementia Diagnosed According to the DSM IV (Diagnostic of Dementia)
Description: The Diagnostic and Statistical Manual of Mental Disorders: 4th Edition of the American Psychiatric Association (DSM-IV, 1994) also outlines diagnostic criteria for dementia of the Alzheimer's type that are generally consistent with the NINCDS-ADRDA criteria.
  National Institute of Neurological and Communicative Diseases and Stroke / Alzheimer's Disease and Related Disorders Association (NINCDS/ADRDA)
Time Frame: At Month 9
Population: ITT population. N=Number of subjects with assessment
Measure: Number; unit: participants
Arm/Group | EGb 120 mg (Open Phase - CNE) | EGb 120 mg (Open Phase - MC)
Number analyzed (Participants) | 21 | 20
participants | 0 | 1

14. Secondary Outcome: Number of Subjects Conversion to Alzheimer's Dementia Diagnosed According to NINCDS-ADRDA (Diagnostic of Alzheimer's)
Description: The most widely accepted diagnostic criteria for probable AD are those offered by the National Institute of Neurological and Communicative Disorders and Stroke and by the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA; McKhann et al., 1984). These criteria include the presence of dementia established by clinical examination and confirmed by neuropsychological testing. The dementia is described as involving multiple, progressive cognitive deficits in older persons in the absence of disturbances of consciousness, presence of psychoactive substances, or any other medical, neurological, or psychiatric conditions that might in and of themselves account for these progressive deficits.
Time Frame: At Month 9
Population: ITT population. N=Number of subjects with assessment.
Measure: Number; unit: participants
Arm/Group | EGb 120 mg (Open Phase - CNE) | EGb 120 mg (Open Phase - MC)
Number analyzed (Participants) | 21 | 20
participants | 0 | 1

15. Secondary Outcome: Change in Cognitive Tests-CDR Score in MC and CNE Groups
Description: as for outcome 2
Time Frame: From Baseline (Month 0) to Month 18
Population: ITT population. N=Number of subjects with assessment.
Measure: Median (Full Range); unit: CDR overall score
Arm/Group | EGb 120 mg (Open Phase - CNE) | EGb 120 mg (Open Phase - MC)
Number analyzed (Participants) | 19 | 12
CDR overall score | 0.00 [0.0 to 0.5] | 0.00 [-0.5 to 0.0]

16. Secondary Outcome: Change in Cognitive Tests-GDS Score in MC and CNE Groups
Description: as for outcome 3
Time Frame: From Baseline (Month 0) to Month 18
Population: ITT population. N=Number of subjects with assessment.
Measure: Median (Full Range); unit: GDS Score
Arm/Group | EGb 120 mg (Open Phase - CNE) | EGb 120 mg (Open Phase - MC)
Number analyzed (Participants) | 19 | 12
GDS Score | 1.00 [-7.0 to 17.0] | 0.50 [-5.0 to 7.0]

17. Secondary Outcome: Change in Cognitive Tests-Verbal Fluency in MC and CNE Groups
Description: as for outcome 4
Time Frame: From Baseline (Month 0) to Month 18
Population: ITT population. N=Number of subjects with assessment.
Measure: Median (Full Range); unit: Number of good answers
Arm/Group | EGb 120 mg (Open Phase - CNE) | EGb 120 mg (Open Phase - MC)
Number analyzed (Participants) | 19 | 12
Number of good answers
  categorical verbal fluency | -1.00 [-18.0 to 20.0] | 1.00 [-9.0 to 10.0]
  lexical verbal fluency | -1.00 [-16.0 to 18.0] | 1.50 [-7.0 to 22.0]

18. Secondary Outcome: Change in Cognitive Tests-MMSE Score in MC and CNE Groups
Description: as for outcome 6
Time Frame: From Baseline (Month 0) to Month 18
Population: ITT population. N=Number of subjects with assessment.
Measure: Median (Full Range); unit: MMSE Score
Arm/Group | EGb 120 mg (Open Phase - CNE) | EGb 120 mg (Open Phase - MC)
Number analyzed (Participants) | 19 | 12
MMSE Score | 0.00 [-4.0 to 2.0] | 0.00 [-5.0 to 4.00]

19. Secondary Outcome: Change in Cognitive Tests-Clock Drawing Test Score in MC and CNE Groups
Description: as for outcome 7
Time Frame: From Baseline (Month 0) to Month 18
Population: ITT population. N=Number of subjects with assessment.
Measure: Median (Full Range); unit: Clock drawing test score
Arm/Group | EGb 120 mg (Open Phase - CNE) | EGb 120 mg (Open Phase - MC)
Number analyzed (Participants) | 19 | 12
Clock drawing test score | 0.00 [-4.0 to 1.0] | 0.00 [-3.0 to 2.0]

20. Secondary Outcome: Change in Cognitive Tests-Cube Drawing Test Score in MC and CNE Groups
Description: as for outcome 8
Time Frame: From Baseline (Month 0) to Month 18
Population: ITT population. N=Number of subjects with assessment.
Measure: Median (Full Range); unit: Cube drawing test score
Arm/Group | EGb 120 mg (Open Phase - CNE) | EGb 120 mg (Open Phase - MC)
Number analyzed (Participants) | 19 | 12
Cube drawing test score | 0.00 [-6.0 to 2.0] | 0.00 [-4.0 to 2.0]

21. Secondary Outcome: Change in Cognitive Tests in MC and CNE Groups - Total Immediate Recall and Delayed Recall Scores of FCSRT
Description: as for outcome 9
Time Frame: From Baseline (Month 0) to Month 18
Population: ITT population. N=Number of subjects with assessment.
Measure: Median (Full Range); unit: Recall score
Arm/Group | EGb 120 mg (Open Phase - CNE) | EGb 120 mg (Open Phase - MC)
Number analyzed (Participants) | 19 | 12
Recall score
  Total Immediate Recall Score of FCSRT | 2.00 [-3.0 to 16.0] | 1.50 [-4.0 to 8.0]
  Total Delayed Recall Score of FCSRT | 0.00 [-6.0 to 6.0] | 0.00 [-2.0 to 2.0]

22. Secondary Outcome: Change in Cognitive Tests-Age-Adjusted Logical Memory (MEM III) in MC and CNE Groups
Description: as for outcome 10
Time Frame: From Baseline (Month 0) to Month 18
Population: ITT population. N=Number of subjects with assessment.
Measure: Median (Full Range); unit: Age adjusted score
Arm/Group | EGb 120 mg (Open Phase - CNE) | EGb 120 mg (Open Phase - MC)
Number analyzed (Participants) | 19 | 11
Age adjusted score | 0.00 [-4.0 to 7.0] | 0.00 [-4.0 to 9.0]

23. Secondary Outcome: Change in Cognitive Tests-Age-Adjusted WAIS in MC and CNE Groups
Description: as for outcome 11
Time Frame: From Baseline (Month 0) to Month 18
Population: ITT population. N=Number of subjects with assessment.
Measure: Median (Full Range); unit: Age adjusted score
Arm/Group | EGb 120 mg (Open Phase - CNE) | EGb 120 mg (Open Phase - MC)
Number analyzed (Participants) | 19 | 12
Age adjusted score | 1.00 [-3.0 to 4.0] | 1.50 [-2.0 to 5.0]

24. Secondary Outcome: Change in Cognitive Tests-Time to Perform TMT in MC and CNE Groups
Description: TMT is a neuropsychological test of visual attention and task switching. The task requires a subject to 'connect-the-dots' of 25 consecutive numbers (1,2,3,etc.) on a sheet of paper or computer screen. The goal of the subject is to finish the test as quickly as possible and the time taken to complete the test is used as the primary performance metric (in seconds). The maximum time allowed is 300 seconds. A negative change score indicates improvement.
  First, in the TMT A, the subject has to connect numbers increasingly as fast as possible.The TMT B requires the subject to connect and letters in an alternating pattern (1-A-2-B-3-C, etc.) in as little time as possible.
Time Frame: From Baseline (Month 0) to Month 18
Population: ITT population. N=Number of subjects with assessment.
Measure: Median (Full Range); unit: Seconds
Arm/Group | EGb 120 mg (Open Phase - CNE) | EGb 120 mg (Open Phase - MC)
Number analyzed (Participants) | 21 | 20
Seconds
  Task A (N=18,12) | -3.00 [-59.0 to 8.0] | -1.00 [-31.0 to 29.0]
  Task B (N=18,11) | -4.50 [-213.0 to 29.0] | -9.00 [-76.0 to 100.0]

25. Secondary Outcome: Number of Subjects Conversion to Alzheimer's Dementia Diagnosed According to the DSM IV (Diagnostic of Dementia)
Description: The Diagnostic and Statistical Manual of Mental Disorders: 4th Edition of the American Psychiatric Association (DSM-IV, 1994) also outlines diagnostic criteria for dementia of the Alzheimer's type that are generally consistent with the NINCDS-ADRDA criteria.
Time Frame: At Month 18
Population: ITT population. N=Number of subjects with assessment.
Measure: Number; unit: participants
Arm/Group | EGb 120 mg (Open Phase - CNE) | EGb 120 mg (Open Phase - MC)
Number analyzed (Participants) | 21 | 20
participants | 0 | 0

26. Secondary Outcome: Number of Subjects Conversion to Alzheimer's Dementia Diagnosed According to NINCDS-ADRDA (Diagnostic of Alzheimer's)
Description: as for outcome 14
Time Frame: At Month 18
Population: ITT population. N=Number of subjects with assessment.
Measure: Number; unit: participants
Arm/Group | EGb 120 mg (Open Phase - CNE) | EGb 120 mg (Open Phase - MC)
Number analyzed (Participants) | 21 | 20
participants | 0 | 0

27. Secondary Outcome: Incidence of Adverse Events (AEs)
Description: The relationship of an adverse event to the study medication will be classified according to the following criteria:
  Related : reports including good reasons and sufficient information (e.g. temporal relationship, dose-response relationship, pharmacology, positive de-challenge and/or re-challenge) to assume a causal relationship with the study drug in the sense that it is plausible, conceivable, or likely
  Not related: reports including good reasons and sufficient information (e.g. no temporal relationship and/or attributable to concurrent disease or other drugs) to rule out a causal relationship with the study drug.
Time Frame: Up to Month 18
Population: Safety population. CNE patients withdrew during the double-blind phase and were also not included in the safety population for open phase (17 months).
Measure: Number; unit: participants
Groups:
- EGb761 120 mg (Double-blind Phase): EGb761 120 mg twice a day for 4 weeks (double-blind phase) for CNE, MC and AD patients
- Placebo (Double-blind Phase): Placebo 1 tablet twice a day for 4 weeks (double-blind phase) for CNE, MC and AD patients
- EGb761 120 mg (Open Phase): EGb761 120 mg twice a day for 17 months (open phase) for MC and CNE patients
Arm/Group | EGb761 120 mg (Double-blind Phase) | Placebo (Double-blind Phase) | EGb761 120 mg (Open Phase)
Number analyzed (Participants) | 23 | 26 | 41
participants
  Any Adverse Events | 5 | 9 | 25
  Any Treatment Emergent | 5 | 8 | 25
  Intensity of Severe Treatment Emergent AEs (TEAEs) | 1 | 0 | 6
  Intensity of moderate TEAEs | 2 | 4 | 14
  Intensity of mild TEAEs | 4 | 5 | 20
  Causality of Related TEAEs | 1 | 2 | 3
  Causality of Non Related TEAEs | 4 | 6 | 25
  Causality and Intensity | 0 | 0 | 0
  At least one related & severe | 0 | 0 | 0
  At least one related & moderate | 0 | 1 | 1
  At least one related & mild | 1 | 2 | 2
  At least one not related & severe | 1 | 0 | 6
  At least one not related & moderate | 2 | 3 | 14
  At least one not related & mild | 3 | 3 | 20
  TEAEs leading to withdrawal | 1 | 2 | 4
  TEAES Leading to Death | 0 | 0 | 0
  Serious AEs (SAEs) | 1 | 0 | 6
  Non SAEs | 5 | 9 | 23

28. Secondary Outcome: Change in Brain Morphology in the MC and CNE Groups as Determined by the Change in Voxel Size
Description: Evolution of brain morphology (degree of cortical atrophy) after 18 months with EGb761, using MRI voxel based morphometry
Time Frame: From Baseline (Month 0) to Month 18
Population: ITT population.
Measure: Median (Full Range); unit: mm3
Groups:
- EGb761 120 mg (CNE): EGb761 120 mg tablet twice a day for 17 months (open phase) for CNE patients
- EGb761 120 mg (MC): EGb761 120 mg 17 months (open phase) for MC patients
Arm/Group | EGb761 120 mg (CNE) | EGb761 120 mg (MC)
Number analyzed (Participants) | 21 | 20
mm3
  Cerebellum | 6454.00 [-42470.0 to 30372.0] | 6168.50 [-38855.2 to 65345.0]
  Left cerebral cortex | 5765.50 [-52347.0 to 97071.0] | 32428.00 [-103527 to 88300.0]
  Left thalamus | 145.20 [-418.9 to 1023.1] | 24.57 [-794.8 to 780.4]
  Left caudate nucleus | 154.68 [-387.3 to 1105.3] | 140.97 [-827.2 to 1384.0]
  Left putamen nucleus | -17.14 [-346.4 to 676.4] | 4.00 [-842.6 to 481.0]
  Left ventral striatum | 65.26 [-99.0 to 157.6] | 81.56 [-57.4 to 236.4]
  Left globus pallidus | 104.75 [-86.2 to 380.4] | 50.66 [-208.7 to 431.8]
  Right cerebral cortex | 5853.00 [-40148.0 to 103200.0] | 38955.50 [-102169 to 97667.0]
  Right thalamus | 144.83 [-715.7 to 669.6] | 14.90 [-570.1 to 755.1]
  Right caudate nucleus | 228.74 [-274.2 to 519.6] | 303.66 [-223.5 to 1084.4]
  Right putamen nucleus | 8.36 [-229.6 to 663.8] | -78.94 [-520.5 to 343.9]
  Right ventral striatum | 65.15 [-5.5 to 198.8] | 70.85 [-13.0 to 287.7]
  Right globus pallidus | 84.68 [-293.0 to 312.6] | 64.82 [-119.3 to 318.8]

ADVERSE EVENTS:
Time Frame: Up to month 18 follow up
Groups:
- EGb761 120 mg (Double-blind Phase): EGb761 120 mg tablet twice a day for 4 weeks (double-blind phase) for CNE, MC, and AD patients
- Placebo (Double-blind Phase): Placebo 1 tablet twice a day for 4 weeks (double-blind phase) for CNE, MC, and AD patients
- EGb761 120 mg (Open Phase): EGb761 120 mg tablet twice a day for 17 months (open phase) for MC and CNE patients
Arm/Group | EGb761 120 mg (Double-blind Phase) | Placebo (Double-blind Phase) | EGb761 120 mg (Open Phase)
Serious Adverse Events (participants affected / at risk) | 1/23 | 0/26 | 6/41
Other Adverse Events (participants affected / at risk) | 5/23 | 9/26 | 23/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EGb761 120 mg (Double-blind Phase) (N=23) | Placebo (Double-blind Phase) (N=26) | EGb761 120 mg (Open Phase) (N=41)
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1
Subclavian artery stenosis (Vascular disorders) | 0 | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EGb761 120 mg (Double-blind Phase) (N=23) | Placebo (Double-blind Phase) (N=26) | EGb761 120 mg (Open Phase) (N=41)
Constipation (Gastrointestinal disorders) | 0 | 0 | 3
Gastro esophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 2
Aerophagia (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Dementia Alzheimer's type (Nervous system disorders) | 0 | 1 | 2
Headache (Nervous system disorders) | 1 | 0 | 1
Essential Tremor (Nervous system disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Hemicephalalgia (Nervous system disorders) | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1 | 1
Syncope vasovagal (Nervous system disorders) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 2
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1
Ear infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 1
Tracheobronchitis (Infections and infestations) | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 3
Insomnia (Psychiatric disorders) | 0 | 0 | 3
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 5
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 2
Macular degeneration (Eye disorders) | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No